CLINICAL TRIAL: NCT02936856
Title: Hepatic Arteriography in Liver Cancer Diagnosis and Staging Applications
Acronym: RDSA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, TaoBai, Researcher, Guangxi Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GuangxiMUBT
Record Dates: First submitted 2016-05-10; First posted 2016-10-18 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: HepatoCellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

ARMS (2):
- After Hepatic Arteriography (Experimental)
  Interventions: Device: Hepatic Arteriography
- Before Hepatic Arteriography (Active Comparator)
  Interventions: Device: Hepatic Arteriography

INTERVENTIONS:
Device: Hepatic Arteriography

SUMMARY:
Primary liver cancer is one of the most common malignant tumor and leading cause of cancer-related death worldwide. Basically therapeutic strategies were considered and given based on the staging of liver cancer. Thus, the confirmatory diagnosis of numbers and distribution of malignant lesions were extreme important. Enhanced CT or MRI is routinely imaging scans to detect and identify lesions. Unfortunately, some malignant lesions usually presented untypical imaging characteristics, especially among lesions no larger than 1 cm, which misleading to the exact staging of liver cancer and the optimal therapeutic strategies.

Basically most of blood supply for malignant liver tumors is from the hepatic artery. Based on this fact, hepatic arterial digital subtraction angiography could potentially elevate the accuracy and sensitivity of detection malignant lesions numbers and distribution.

In this study the investigators will compare the numbers and distribution of malignant lesions before and after hepatic arteriography, then to revise the staging of liver cancer and to provide better therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary liver cancer who is firstly diagnosed in Affiliated Tumor Hospital of Guangxi Medical University after November 2015, and the clinical diagnostic criteria is according to China's "primary liver cancer diagnostic and treatment practices (2011)". Clinical diagnostic criteria: In all solid tumors, there is only hepatocellular carcinoma can use clinical diagnostic criteria, which is recognized by domestic and foreign countries. Combined with China's national conditions, history of the national standards and clinical practice, the Expert Group can establish the clinical diagnosis of hepatocellular carcinoma requested the following conditions 1 + 2a or 1 + 2b + 3 at the same time satisfy:

  * Patients have evidence of liver cirrhosis or HBV and / or HCV infection (HBV and / or HCV antigen positive).
  * Typical imaging features of hepatocellular carcinoma: liver lesion shows arterial hypervascularity and venous or delayed phase washout in multidetector CT scan and / or dynamic contrast enhanced MRI. a: If the liver lesion diameter≥2cm, the diagnosis of hepatocellular carcinoma can be made when typical imaging features show in one of the imaging methods. b: If the liver lesion diameter is between 1 to 2cm, the diagnosis of hepatocellular carcinoma can be made when typical imaging features show in both of the imaging methods.
  * Serum AFP≥400μg/L for 1 month or ≥200μg/L for 2 month, and can rule out other causes of AFP increasing (pregnancy, reproductive system embryo-derived tumors, active liver disease and secondary liver cancer, etc.).

Exclusion Criteria:

* Patients do not conform to China's "primary liver cancer diagnostic and treatment practices (2011)".
* Patients allergic to Iodine-containing contrast agents or with obvious hyperthyroidism.
* Patients with severe cardiovascular disease or liver or renal insufficiency, who do not tolerate digital subtraction angiography or will significantly increase the risk of diseases.
* Patients have severe coagulation disorders or are extreme weak.
* Patients have fever or have infection on the puncture site.
* Patients suffer from mental illness or cannot cooperate with the treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Detection of numbers of confirmatory diagnosis of malignant lesions before and after hepatic arteriography | 1 year
  Comparing the numbers and distribution of confirmatory diagnosis (positive/negative) of malignant lesions before and after hepatic arteriography, which to re-evaluate the staging of primary liver cancer and to further provide better therapeutic strategies

SECONDARY OUTCOMES:
Detection of distribution of confirmatory diagnosis of malignant lesions before and after hepatic arteriography | 1 year
  Comparing the distribution of confirmatory diagnosis (positive/negative) of malignant lesions before and after hepatic arteriography, which to re-evaluate the staging of primary liver cancer and to further provide better therapeutic strategies

CONTACTS AND LOCATIONS:
Locations (1):
- TaoBai, Nanning, Guangxi, China